CLINICAL TRIAL: NCT07096765
Title: Effect of Injection Duration of Fascial Plane Blocks on Block Success and Postoperative Analgesia in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Effect of Injection Duration of Fascial Plane Blocks on Block Success
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Korgün Ökmen, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2024-ТВЕK 2025/07-05
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Nerve Block
MeSH Terms: interventions — O-antigen, Acinetobacter strain 90; Sensitivity Training Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional (Active Comparator): During the fascia block application, the injection will be administered using the conventional method without any specific time limit.
  Interventions: Drug: Group C
- One-minute injection (Active Comparator): During the fascia block application, the injection will be administered within 1 minute.
  Interventions: Drug: Group O
- Two-minute injection (Active Comparator): During the fascia block application, the injection will be administered within 2 minutes.
  Interventions: Drug: Group T

INTERVENTIONS:
Drug: Group O — Ultrasound guided External Oblique And Rectus Abdominis Plane (EXORA) Block block (0.3 ml/kg ,
  %0.25 bupivacaine) will be performed Drug: Tramadol 400 mg tramadol, IV 4 mg/ mL tramadol solution into 100 mL normal saline; Patient-controlled analgesia settings: 0.3 mg/kg bolus, 10 mg Demand dose and 20 min lock out interval, six-hour limit infusion to attain 100 mg. Maximum daily dose was set at 400 mg.
  Arms: One-minute injection
Drug: Group T — Ultrasound guided External Oblique And Rectus Abdominis Plane (EXORA) Block block (0.3 ml/kg ,
  %0.25 bupivacaine) will be performed Drug: Tramadol 400 mg tramadol, IV 4 mg/ mL tramadol solution into 100 mL normal saline; Patient-controlled analgesia settings: 0.3 mg/kg bolus, 10 mg Demand dose and 20 min lock out interval, six-hour limit infusion to attain 100 mg. Maximum daily dose was set at 400 mg.
  Arms: Two-minute injection
Drug: Group C — Ultrasound guided External Oblique And Rectus Abdominis Plane (EXORA) Block block (0.3 ml/kg ,
  %0.25 bupivacaine) will be performed Drug: Tramadol 400 mg tramadol, IV 4 mg/ mL tramadol solution into 100 mL normal saline; Patient-controlled analgesia settings: 0.3 mg/kg bolus, 10 mg Demand dose and 20 min lock out interval, six-hour limit infusion to attain 100 mg. Maximum daily dose was set at 400 mg.
  Arms: Conventional

SUMMARY:
This prospective observational study aims to evaluate the impact of injection duration during fascial plane blocks on block success and analgesic efficacy in patients undergoing laparoscopic cholecystectomy. The hypothesis is that shorter injection durations increase injection pressure, potentially limiting local anesthetic spread, while longer durations facilitate broader anesthetic distribution.

DETAILED DESCRIPTION:
Fascial plane blocks involve injecting local anesthetics between two anatomical fascial layers, with analgesia achieved by anesthetic diffusion through the fascial plane. However, anesthetic spread may vary significantly based on injection technique, speed, and pressure. This study hypothesizes that injection duration directly influences injection pressure, local anesthetic distribution, and consequently, the extent of sensory blockade and analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic cholecystectomy surgery
* Patients with ASA (American Society of Anaesthetists) scores I and III will be included.

Exclusion Criteria:

* Uncontrolled Arterial Hypertension
* Uncontrolled Diabetes Mellitus,
* Mental retardation
* Antidepressant use
* Metabolic disorders
* Bleeding diathesis
* Patients with a body mass index above 30

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
sensory block distribution | Postoperative 24 hours
  The distribution of sensory block will be evaluated using pinprick and cold tests at 2, 6, 12 and 24 hours after surgery.
  With the pinprick, the gently touches the skin with the pin or back end and asks the patient whether it feels sharp or blunt.

SECONDARY OUTCOMES:
NRS | Postoperative 24 hours
  The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
tramadol consumption | Postoperative 24 hours]
Pressure values | During the procedure
  Pressure values (mm/hg) measured using the infusion device during block application.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No